CLINICAL TRIAL: NCT01246414
Title: Inflammatory Markers in Exhaled Breath Condensates From Asthmatic Patients
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Jettanong Klaewsongkram, MD., Chulalongkorn University
Other Study IDs: Chula-ARC 001/10
Record Dates: First submitted 2010-01-04; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: Asthma; Exhaled breath condensates; Cytokines
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Exhaled breathe condensates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Allergic asthma: Patients with allergic asthma
- Non-allergic asthma: Patients with non-allergic asthma
- Non-asthmatic controls: Non-asthmatic controls

SUMMARY:
This study aims to compare the inflammatory mediators in exhaled breathe condensates from allergic and non-allergic asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed as asthma at least 6 months before enrolled to the study
2. Known skin prick test results to aeroallergens ; either positive or negative
3. 15-65 years of age

Exclusion Criteria:

1. On oral or inhaled corticosteroids within 1 month before the study
2. Having asthma exacerbation
3. Being pregnant
4. Suffering from severe systemic disease/ in bad health

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Asthmatic patients in Allergy clinic, King Chulalongkorn Memorial Hospital (10 allergic and 10 non-allergic) and 10 non-asthmatic controls will be enrolled to this study to collect exhaled breathe condensates (EBC) and measure levels of inflammatory cytokines in EBC
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Levels of inflammatory cytokines in exhaled breathe condensates | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Boonpiyathad S, Pornsuriyasak P, Buranapraditkun S, Klaewsongkram J. Interleukin-2 levels in exhaled breath condensates, asthma severity, and asthma control in nonallergic asthma. Allergy Asthma Proc. 2013 Sep-Oct;34(5):e35-41. doi: 10.2500/aap.2013.34.3680. PMID 23998235